CLINICAL TRIAL: NCT07244458
Title: Dietary Peanut Intake and Nutrition-Related Outcomes in Individuals Using GLP-1 Receptor Agonists: A Randomized Controlled Trial
Brief Title: Dietary Peanuts and Nutrition-Related Outcomes
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ian J. Neeland, MD (Other)
Responsible Party: Sponsor-Investigator, Ian J. Neeland, MD, Director, UH Center for Cardiovascular Prevention, University Hospitals Cleveland Medical Center
Organization: University Hospitals Cleveland Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: STUDY20250426
Record Dates: First submitted 2025-11-17; First posted 2025-11-24 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Dietary Change; Obesity & Overweight; Food Acceptance
Keywords: Dietary quality; Eating enjoyment; Satiety; Weight-related outcomes
MeSH Terms: conditions — Obesity; Overweight | interventions — Absorptiometry, Photon

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Peanut Group (Experimental): Participants in this group will eat 2 ounces, or 53 grams of dry-roasted, lightly salted (low sodium) each day along with their regular diet.
  Interventions: Dietary Supplement: Peanuts; Procedure: Dual-energy X-ray absorptiometry (DEXA) scans
- No Peanut Group (Active Comparator): Participants in this group will continue eating regular diet without peanuts.
  Interventions: Procedure: Dual-energy X-ray absorptiometry (DEXA) scans

INTERVENTIONS:
Dietary Supplement: Peanuts — Participants will eat 2 ounces, or about 53 grams, of dry-roasted, lightly salted peanuts each day along with their regular diet
  Arms: Peanut Group
Procedure: Dual-energy X-ray absorptiometry (DEXA) scans — DEXA scans will be used to measure body fat

SUMMARY:
This study will look at how eating peanuts every day might affect participants weight, how healthy their diet is, and how they feel when eating. Investigators want to see if adding peanuts to meals for 12 weeks helps participants feel fuller, have more energy, and improve body composition. The study will include adults who have been taking GLP-1 medicines like semaglutide or tirzepatide for at least three months. Investigators also want to see if eating peanuts improves overall diet quality and health markers like tiredness and certain levels in blood.

ELIGIBILITY:
Inclusion Criteria:

* Individuals with a BMI ≥30 kg/m2 who intend to be continuously using semaglutide or tirzepatide for a clinical indication and remain on the therapy for at least 6 months

Exclusion Criteria:

* No use or contraindication to use of a GLP-1 RA
* Known allergy to nuts
* Pregnant or breastfeeding
* Incarcerated

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Change is Satiety as measured by the Hunger and Satiety Visual Analog Scales (VAS) | Baseline, End of study (12 weeks)
  Participants will rate their perceived hunger, fullness, and desire to eat on a 100-mm scale, with endpoints ranging from "not at all" to "extremely" for each category.
Change in fatigue as measured by the Fatigue Severity VAS-F Survey | Baseline, End of study (12 weeks)
  Each item is presented on a 100-mm scale, with endpoints labeled to reflect the extremes of the sensation being measured (e.g., "Not at all tired" to "Extremely tired"). Participants will complete the VAS-F at consistent times of the day to minimize variability. Scores will be recorded both before and after meals to capture potential fluctuations in energy levels.
Change in mood/well-being as measured by the Mental clarity, energy levels, and motivation VAS. | Baseline, End of study (12 weeks)
  Each item is presented on a 100-mm scale, with endpoints labeled to reflect the extremes of being measured ranging from, for example, "not at all" to "extremely".
Change in dietary quality as measured by Healthy Eating Index (HEI) | Baseline, End of study (12 weeks)
  HEI scores measure how well a diet aligns with the Dietary Guidelines for Americans. The scores range from 0 to 100, with higher scores indicating foods align with key dietary recommendations and dietary patterns published in the Dietary Guidelines.
Change in food enjoyment as measured by the Food Pleasure Scale (FPS) | Baseline, End of study (12 weeks)
  The FPS is a validated 21-item tool designed to measure multiple dimensions of food-related enjoyment, including sensory characteristics (appearance, odor, taste, texture), expectations and desires (memories, habits, expectations, choices, needs), and other relevant factors. The importance of each item in relation to general pleasurable experiences of food is rated on a 5-point ordinal scale ranging from 1 ("Not important at all") to 5 ("Extremely important").
Change in fasting glucose as measured by medical record review | Baseline, End of study (12 weeks)
Change in HbA1c as measured by medical record review | Baseline, End of study (12 weeks)
Change in total cholesterol as measured by medical record review | Baseline, End of study (12 weeks)
Change in LDL-C as measured by medical record review | Baseline, End of study (12 weeks)
Change in HDL-C as measured by medical record review | Baseline, End of study (12 weeks)
Change in triglycerides as measured by medical record review | Baseline, End of study (12 weeks)
Change in physical activity as measured by International Physical Activity Questionnaire (IPAQ) | Baseline, End of study (12 weeks)
  The IPAQ short form consists of 7 questions designed to assess physical activity levels over the past 7 days in adults. The score is calculated using published guidelines and ranges from 0 to infinity and measures physical activity in median median MET-minutes/week. This is a continuous measure and is calculated as: Total MET-min/week = (Walk METs*min*days) + (Moderate activity METs*min*days) + Vigorous activity METs*min*days).

SECONDARY OUTCOMES:
Change in body weight as measured by medical record review | Baseline, End of study (12 weeks)
Change in waist circumference as measured by medical record review | Baseline, End of study (12 weeks)
Change in hip circumference as measured by medical record review | Baseline, End of study (12 weeks)
Change in fat mass as measured by DEXA scan | Baseline, End of study (12 weeks)
Change in lean body mass as measured by DEXA scan | Baseline, End of study (12 weeks)
Change in overall body fat percentage as measured by DEXA scan | Baseline, End of study (12 weeks)

CONTACTS AND LOCATIONS:
Overall Officials: Ian Neeland, MD, Principal Investigator — University Hospitals Cleveland Medical Center; Abigail Raffner, MD, Principal Investigator — University Hospitals Cleveland Medical Center
Locations (1):
- University Hospitals Cleveland Medical Center, Clevland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No